CLINICAL TRIAL: NCT04894747
Title: Comparing Postprandial Muscle Protein Synthesis Rates Following the Consumption of Mycoprotein, Pea Protein and a Mycoprotein/Pea Protein Blend in Resistance Trained Individuals
Brief Title: Mycoprotein and Pea Protein Blend and Muscle Protein Synthetic Response
Acronym: BPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Quorn (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 200325_B_04UOE
Record Dates: First submitted 2021-05-05; First posted 2021-05-20 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Muscle Protein Synthesis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mycoprotein (Experimental): Bolus ingestion of mycoprotein providing 25g of protein.
  Interventions: Dietary Supplement: Bolus ingestion of protein
- Pea protein (Experimental): Bolus ingestion of pea protein providing 25g of protein.
  Interventions: Dietary Supplement: Bolus ingestion of protein
- Mycoprotein/pea protein dry blend (Experimental): Bolus ingestion of mycoprotein/pea protein dry blend providing 25g of protein.
  Interventions: Dietary Supplement: Bolus ingestion of protein

INTERVENTIONS:
Dietary Supplement: Bolus ingestion of protein — Ingestion of 25g of protein
  Other Names: Protein ingestion

SUMMARY:
Dietary protein is vital for the preservation of health and optimal adaptation to training. Plant proteins are considered inferior to animal proteins with respect to their ability to stimulate an acute muscle building response and therefore support long-term muscle reconditioning. Pea protein is a highly commercially available plant proteins source (available as supplements, food ingredients etc.), yet there is no research investigating its ability to stimulate a muscle building response. The investigators aim to assess the effect of consuming pea protein on muscle protein synthesis rates and compare these results to mycoprotein, a source known to elicit a robust anabolic response.

Pea protein is lower in some of the essential amino acids, namely methionine, which could mean it is less effective compared with mycoprotein which has a more complete amino acid profile. So in addition to comparing pea with mycoprotein, the investigators also want to compare to a blend of pea and mycoprotein to see if replenishing the amino acid content in pea 'rescues' the anabolic response.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30
* Resistance trained

Exclusion Criteria:

* Any metabolic impairment
* Smoking
* Use of over the counter pharmaceuticals (excluding oral contraceptives and contraceptive devices).
* A personal family history of epilepsy, seizures or schizophrenia.
* Allergic to Quorn/mycoprotein/edible fungi/environmental mould products.
* Any motor disorder.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 8.5 hours
  The rate of synthesis of new muscle protein (Fractional synthetic rate %/h)

SECONDARY OUTCOMES:
Plasma amino acid kinetics | 8.5 hours
  The appearance of amino acids from the protein drink in the circulation.
Serum insulin concentrations | 8.5 hours
  Basal and postprandial concentrations of serum insulin
Translocation of mTOR via immunohistochemistry | 8.5 hours
  Locality of mTOR within the muscle cell
mTOR phosphorylation via ATP kinase assay | 8.5 hours
  The amount of mTOR that has been activated in the muscle cell

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No